CLINICAL TRIAL: NCT05457049
Title: Dynamic Observational Strategy for Stage IB-IIIA Non-Small Cell Lung Cancer Patients After Complete Resection Based on Longitudinal Undetectable Molecular Residual Disease: Prospective, Multicenter, Single-Arm Study
Brief Title: Adjuvant Therapy Omission for Resected NSCLC Patients With Longitudinal Undetectable MRD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Principal Investigator, Guangdong Association of Clinical Trials
Other Study IDs: CTONG 2201
Record Dates: First submitted 2022-07-09; First posted 2022-07-13 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Molecular residual disease; Adjuvant therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Every MRD test will take 20ml peripheral blood for DNA extraction.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Undetectable MRD: Stage IB-IIIA NSCLC patients who after complete resection. And patients who maintain MRD negativity in two-round MRD landmark test (first in 3-7 days after surgery, second in 1 months ±7 days after surgery) will be enrolled. And patients will be under close dynamic monitoring at least two years.
  Interventions: Diagnostic Test: Molecular residual disease test

INTERVENTIONS:
Diagnostic Test: Molecular residual disease test — OncoMRD Lung

SUMMARY:
Molecular residual disease (MRD) has strong relationship with clinical outcome in multiple solid tumors. Here, the investigators try to verify the negative predictive value of undetectable MRD, which is considered as a superior prognostic factor for resected NSCLC patients, and not requiring excessive adjuvant therapy. Stage IB-IIIA resected NSCLC patients with landmark and longitudinal undetectable MRD are enrolled and under close surveillance in this study.

DETAILED DESCRIPTION:
Stage IB-IIIA resected NSCLC patients will undergo two-round MRD tests after operation, first in 3-7 days and second in 1 month after operation. And patients who confirm two-round landmark undetectable MRD will be enrolled. Enrolled patients will be under close MRD and imaging monitoring without any adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Stage IB-IIIA non-small cell cancer patients who after complete resection.
* ≥18 years.
* Two-round MRD tests confirm landmark undetectable MRD.
* Expected survival ≥12 weeks.
* Expected survival ≥12 weeks.
* ECOG PS 1-2.
* Willing to accept MRD monitoring every 3 months for a total of 2 years after operation.

Exclusion Criteria:

* Patients who had previously undergone radiotherapy or chemotherapy or any other anti-tumor therapy.
* Patients with a history of other malignancies in the past 5 years.
* Any unstable systemic disease (eg, active infection, high-risk hypertension, unstable angina, congestive heart failure, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IB-IIIA NSCLC patients who after complete resection and undetectable landmark MRD.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Two-years disease free survival rates for patients with longitudinal undetectable MRD | 2 year
  The 2-year DFS rate of patients who maintain 2-years undetectable MRD.

SECONDARY OUTCOMES:
Two-years disease free survival rates for patients with six months longitudinal undetectable MRD | 2 year
  The 2-year DFS rate of patients who maintain 6-months undetectable MRD.
Two-years disease free survival rates for patients with 12-months longitudinal undetectable MRD | 2 year
  The 2-year DFS rate of patients who maintain 12-months undetectable MRD.
Two-years disease free survival rates for patients with 18-months longitudinal undetectable MRD | 2 year
  The 2-year DFS rate of patients who maintain 18-months undetectable MRD.
Two-years event-free survival rates for enrolled patients in two years | 2 year
  The events are defined as disease recurrence or detectable MRD.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang JT, Liu SY, Gao W, Liu SM, Yan HH, Ji L, Chen Y, Gong Y, Lu HL, Lin JT, Yin K, Jiang BY, Nie Q, Liao RQ, Dong S, Guan Y, Dai P, Zhang XC, Yang JJ, Tu HY, Xia X, Yi X, Zhou Q, Zhong WZ, Yang XN, Wu YL. Longitudinal Undetectable Molecular Residual Disease Defines Potentially Cured Population in Localized Non-Small Cell Lung Cancer. Cancer Discov. 2022 Jul 6;12(7):1690-1701. doi: 10.1158/2159-8290.CD-21-1486. PMID 35543554
- [Derived] Zhang JT, Dong S, Gu WQ, Zhao N, Liang Y, Tang WF, Liu SY, Wang F, Wang GS, Peng B, Wu N, Yan S, Geng GJ, Xie ZF, Yang YL, Zhang JH, Zhang T, Yang N, Jiao WJ, Xiong YY, Cai M, Li F, Chen RR, Yan HH, Maggie Liu SY, Yi X, Zhong WZ, Yang XN, Wu YL. Adjuvant Therapy-Free Strategy for Stage IB to IIIA Non-Small-Cell Lung Cancer Patients After Radical Resection Based on Longitudinal Undetectable Molecular Residual Disease: Prospective, Multicenter, Single-Arm Study (CTONG 2201). Clin Lung Cancer. 2024 Jan;25(1):e1-e4. doi: 10.1016/j.cllc.2023.09.008. Epub 2023 Oct 6. PMID 37880076